CLINICAL TRIAL: NCT04688723
Title: RE-DUAL PCI Real Life Registry Dual Therapy With Dabigatran/Ticagrelor Versus Dual Therapy With Dabigatran/Clopidogrel in ACS Patients With Indication for NOAC Undergoing PCI
Brief Title: Dual Therapy With Dabigatran/Ticagrelor Versus Dual Therapy With Dabigatran/Clopidogrel in ACS Patients With Indication for NOAC Undergoing PCI
Acronym: RE-DUAL PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20200196
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction; Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction; Atrial Fibrillation | interventions — Dabigatran; Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran/Clopidogrel (Active Comparator): Patiënt receive standard care, with dabigatran + clopidogrel 75mg once daily up to 12 months.
  Interventions: Drug: Dabigatran + clopidogrel
- Dabigatran/Ticagrelor (Experimental): Patiënt receive standard care, with dabigatran + ticagrelor 90mg twice daily up to 12 months.
  Interventions: Drug: Dabigatran + Ticagrelor

INTERVENTIONS:
Drug: Dabigatran + Ticagrelor — Patiënt interventional treatment, with dabigatran + ticagrelor (Brilique) 90mg twice daily up to 12 months.
  Arms: Dabigatran/Ticagrelor
Drug: Dabigatran + clopidogrel — Patiënt interventional treatment, with dabigatran + clopidogrel (plavix) 75mg once daily up to 12 months.
  Arms: Dabigatran/Clopidogrel

SUMMARY:
A real world registry to compare dual therapy with Dabigatran/Ticagrelor to dual therapie with Dabigatran/Clopidogrel in patients with an indication for NOAC undergoing PCI in the setting of ACS. Hypothesis: Dual therapy with Dabigatran/Ticagrelor will be non-inferior in reducing the risk of bleeding compared to Dual therapy with Dabigatran/Clopidogrel (RE-DUAL PCI trial based) in patients with an indication for NOAC undergoing PCI in the setting of ACS. Thromboembolic events, stent thrombosis and death will be evaluated for estimation of events between both groups. Data will be pooled for this secondary endpoint with data from the upcoming WOEST-3 trial to compare both treatments.

DETAILED DESCRIPTION:
The REDUAL PCI Registry will we be an open-label multicenter registry based randomised controlled trial (RBRCT) within the ZON-HR collaboration in 4 of the 6 centers in the Netherlands: Maastricht Universitair Medisch Centrum (Maastricht), Zuyderland (Heerlen and Sittard), Vie Curi (Venlo) and Radboud Medisch Centrum (Nijmegen). Isala (Zwolle) and Canisius Wilhelmina ziekenhuis (Nijmegen) will not be part of this study. This study is Investigator initiated with an unrestricted grant from Boehringer Ingelheim (subsidising party). This study is also to be noted as a Post Authorisation Safety Study (PASS). Patients 1000 patients with an indication for NOAC, who underwent successful PCI with Drug Eluting Stent (DES) in the setting of ACS will be included and randomised at each of the 4 centers of the ZON-HR. After randomisation, patients will be treated with Dual therapy with Dabigatran/Clopidogrel or with Dabigatran/ Ticagrelor. A total of 1000 patients in 4 centers will be included: 250 patients in each center. In each center inclusion and randomisation will be executed within 48 hours after PCI. Inclusions are expected to be done within 1 year. After inclusion of the interventional (Dual therapy with Dabigatran/Ticagrelor) and control group (Dual therapy with Dabigatran/Clopidogrel), follow-up of 1 year is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients having an indication for a NOAC or will start with oral anticoagulation (NOAC). Permanent, persistent or paroxysmal atrial fibrillation are eligible.
* PCI and successful stenting with DES for ACS (unstable angina pectoris, NSTEMI, STEMI)
* Written informed consent.

Exclusion Criteria:

* Patients unable or unwilling to comply with the protocol or with life expectancy shorter than the duration of the study
* Glomerular filtration rate < 30 ml/min
* Heart valve prosthesis (mechanical or biological)
* Cardiogenic shock
* Contra-indication for Dabigatran, Ticagrelor or Clopidogrel

  * Liver dysfunction (ALAT, ASAT, Alkaline phosphatase > 3x upper limit of normal) or liver disease (like hepatitis A, B, C)
  * Lesion or condition with a significant risk of serious bleeding, such as; current or recent gastrointestinal ulceration; malignant neoplasms with more bleeding risk; recent brain / spinal cord injury; recent surgery on the brain, spinal cord or eyes; recent or history of intracranial haemorrhage; oesophageal varices; arteriovenous malformations; vascular aneurysms; o severe intraspinal or intracerebral vascular abnormalities.
  * comedication with cyclosporine, itraconazole, ketoconazole (systemic) and glecaprevir / pibrentasvir, dronedarone, rifampicine, carbamazepine, St. Jan's wort or phenytoin o Comedication with tacrolimus is not recommended.
* Allergy to for Dabigatran, Ticagrelor or Clopidogrel
* Pregnancy
* Significant thrombocytopenia (platelet count < 50x10 9/L)
* Major bleeding according to BARC ≥3 within the past 6 months.
* Weight < 50 kg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 12 months
  Bleeding defined as BARC bleeding score ≥2

SECONDARY OUTCOMES:
Myocardial Infarction | 12 months
  Myocardial Infarction
Cerebrovascular accident | 12 months
  Cerebrovascular accident, ischemic of haemorrhagic
Systemic Embolic Complications | 12 months
  Systemic Embolic Complications
Death | 12 months
  Death
Combined endpoint of ischemic events | 12 months
  All secondary outcomes combined into one endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No